CLINICAL TRIAL: NCT03355144
Title: Resident Observed Burnout After Daily Supplementation With Coffee
Acronym: ROBSTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-01011
Record Dates: First submitted 2017-11-22; First posted 2017-11-28 (Actual); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: Burnout, Professional
MeSH Terms: conditions — Burnout, Professional | interventions — Coffee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Internal Medicine residents at NYU (Experimental): effect of supplying Internal Medicine residents at NYU with free coffee on self reported features of psychological health, energy and burnout
  Interventions: Dietary Supplement: Daily Supplementation with Coffee

INTERVENTIONS:
Dietary Supplement: Daily Supplementation with Coffee — At the beginning of study week 2 (study day 8), two coffee machines (one Nespresso Inissia and one Hamilton Beach 46205 12 Cup Programmable Coffee Maker) will be installed in the resident work rooms at each site.
  Subjects will be provided with free coffee beans, milk, cream, sugar and sweetener

SUMMARY:
Coffee drinking is frequently reported as a negative outcome in studies on burnout, but the effect of an increased coffee intake on resident burnout has not been reported in the literature. This study is a prospective, interventional cohort study enrolling up to 50 residents from the Internal Medicine Residency Program to look at the relationship between coffee and resident burnout.

DETAILED DESCRIPTION:
Resident burnout is increasingly being recognized as detrimental to both physician well being and patient care. It has been linked to an increased rate of medical errors and a reduced quality of patient care. In addition, there have been multiple high-profile physician suicides in the past years. This has resulted in a renewed focus on physician mental health and workload.

ELIGIBILITY:
Inclusion Criteria:

* A resident in the NYU Internal Medicine residency program

Exclusion Criteria:

* Allergy or intolerance to coffee or caffeine
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2018-03-22 (Actual); Primary Completion 2018-04-12 (Actual); Study Completion 2018-04-12 (Actual)

PRIMARY OUTCOMES:
Self reported feelings of burnout | 1 Month
  14 question survey measuring number of cups of coffee and level of exhaustion

SECONDARY OUTCOMES:
Coffee consumption measured by self reporting questionaire | 1 Month
  Measured by self reporting questionnaire
Self reported emotional well being | 1 Month
  14 question survey with questions measuring emotional wellbeing
Self reported feelings of value | 1 Month
  14 question survey with questions measuring feelings of self value

CONTACTS AND LOCATIONS:
Overall Officials: Steven Liu, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States